CLINICAL TRIAL: NCT02017353
Title: Effect of Curcumin Addition to Standard Treatment on Tumour-induced Inflammation in Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: Reliable Cancer Therapies (Industry)
Responsible Party: Principal Investigator, Sandra Tuyaerts, PhD, University Hospital, Gasthuisberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S55201; 2013-001737-40 (EudraCT Number)
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Curcuphyt (Experimental): Intake of Curcuphyt capsules, 2 g per day during 2 weeks
  Interventions: Dietary Supplement: Curcuphyt

INTERVENTIONS:
Dietary Supplement: Curcuphyt
  Other Names: Meriva

SUMMARY:
This therapy aims to determine whether curcumin can inhibit tumor induced inflammation in patients with endometrial carcinoma. In addition, curcumin could possibly induce a better functioning of chemotherapy and a decrease in toxicity from chemotherapy. Various studies have demonstrated that curcumin can have an effect on tumor growth and the development of metastases.

DETAILED DESCRIPTION:
Various cancer types are associated with chronic inflammation. During the formation of cancer the immune system is being activated by the tumor in order to evoke an anti-tumor immune response. However, as the tumor develops, this gives rise to a chronic inflammation, causing the immune system to malfunction. This is being highlighted by the fact that different chronic inflammatory diseases are associated with an increased risk of cancer (f.i. chronic inflammatory bowel diseases and colon cancer, prostatitis and prostate cancer, hepatitis and liver cancer). Endometrial cancer reveals different aspects of inflammation, including cytokine secretion and the infiltration of immune cells in this type of tumors. It is presumed that hormonal fluctuations and genetic changes contribute to the formation of a pro-inflammatory environment that stimulates tumor growth. Cancer cells of endometrial tumors do not only produce immunomodulatory mediators, but also attract different sorts of cells of the immune system that stimulate tumor growth.

It has already been demonstrated in mice models and in vitro experiments that curcumin shows strong anti-inflammatory effects that can slow down tumor growth and/or prevent formation of metastases. In addition, it has been noticed in these models that curcumin also has a positive effect on the functioning of various chemotherapeutic drugs, causing their effect to enhance or their toxicity to decrease.

Clinical studies investigating the anti-inflammatory effect of curcumin are rare, but these studies do reveal a suppression of the inflammation. The primary reason why clinical studies with curcumin are rare is because of the bad intake of curcumin in the human body. Recently, there has been a lot of research carried out regarding the development of new formulations of curcumin that lead to a better intake in the human body. The best nutritional supplement containing curcumin that has been developed so far is Meriva®, which is commercialized in Belgium under the name "CurcuPhyt".

ELIGIBILITY:
Inclusion Criteria:

* Endometrial carcinoma at time of recurrence
* No life-threatening metastases

Exclusion Criteria:

* Other active malignancy
* Documented autoimmune disease
* Currently ongoing immunosuppressive therapy
* Simultaneous treatment according to other clinical trials
* Documented immune deficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory markers in peripheral blood from baseline | baseline, day 1, day 7, day 14, day 21

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | up to 3 weeks
Change from Baseline in Quality of Life score | baseline, day 14

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Amant, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospital KU Leuven Campus Gasthuisberg, Leuven, Belgium